CLINICAL TRIAL: NCT01463670
Title: A Phase II Clinical Trial of Lenalidomide Intensification in Patients With Serologic/Asymptomatic Progression of Multiple Myeloma While on Lenalidomide Maintenance
Brief Title: Lenalidomide Intensification in Patients With Serologic/Asymptomatic Progression of Multiple Myeloma While on Lenalidomide Maintenance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Montefiore Medical Center (Other); State University of New York - Downstate Medical Center (Other); University of Rochester (Other); Weill Medical College of Cornell University (Other); Stamford Hospital (Other); Columbia University (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-107
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
Keywords: LENALIDOMIDE (CC-5013); BONE MARROW; 11-107
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

ARMS (1):
- lenalidomide (Experimental): The proposed study is designed as a Phase II, multi-center trial of lenalidomide intensification in patients with asymptomatic POD while on low dose lenalidomide maintenance after HDM/ASCT or on continuous/maintenance therapy after initial treatment.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — patients will begin therapy with lenalidomide 25 mg daily, 21 days out of a 28 day schedule. All patients will be evaluated monthly after every cycle. The dose will be adjusted downward in response to side effects and according to specific guidelines. Symptomatic POD occurring at any time during the study will result in removal of the patient from the study. After 2 cycles of lenalidomide, patients with at least stable disease (SD) will continue lenalidomide indefinitely until asymptomatic POD, at which time dexamethasone will be added at a dose of 40mg weekly. On the other hand, patient with asymptomatic POD after 2 cycles of lenalidomide will have dexamethasone added at a dose of 40 mg weekly. Patients with any type of POD after any cycle that includes dexamethasone will be taken off study. Patients can remain on study on lenalidomide or lenalidomide/dexamethasone indefinitely as long as they do not have POD as stated above and they tolerate the treatment.

SUMMARY:
The purpose of this study is to determine whether this disease will get better if treated with higher doses of Lenalidomide even if the disease returns while taking low doses of Lenalidomide. In patients with multiple myeloma treated with Lenalidomide maintenance, the disease will return. However, the physician currently does not know if the disease would respond to treatment with higher doses of Lenalidomide. This is very important for patients with multiple myeloma because the number of drugs available to treat the disease are limited. It is important to know if Lenalidomide remains still effective and if it can still be used in this situation. This study will try to find out what effects, good and/or bad higher doses of Lenalidomide has on the patient and the disease after it has returned.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or above at the time of enrollment.
* Patients must show evidence of asymptomatic relapse and/or progression of disease (increasing M spike in serum or urine by consensus criteria) while on lenalidomide maintenance after HDM/ASCT as part of initial line of therapy.
* Patients who have not had an HDM/ASCT as part of initial line of therapy but who are on continuous/maintenance lenalidomide after initial therapy will be permitted on study.
* Patient must have myeloma that is measurable by either serum or urine evaluation of the monoclonal component or by assay of serum free light chains. Measurable disease is defined as one or more of the following: serum M-protein ≥ to 0.5 g/dl, urine M-protein ≥ 200 mg/24 h, and/or serum FLC assay: involved FLC level > 10 mg/dL with abnormal serum FLC ratio.
* Patients must have adequate organ function including: Hepatic function with Bilirubin <2x the upper limit of normal and ALT and AST < 3 x the upper limit of normal; renal function with creatinine clearance ≥ 60 ml/min using the Cockcroft-Gault formula; hematologic function as defined by an absolute neutrophil count > 1000 neutrophils per microliter, platelet > 50,000 platelets per microliter and hemoglobin of ≥ 9 gm/dL without transfusion support
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of child bearing potential (FCBP) must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program
* FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

Exclusion Criteria:

* Patients with symptomatic relapse and/or progression of multiple myeloma. (Appendix A).
* Patients with plasma cell leukemia.
* Karnofsky performance score less than 70% or ECOG performance status greater than 2.
* Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms).
* Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ or other cancer treated with curative intent > 5 years previously. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Protocol Chairs.
* Female patients who are pregnant (positive HCG) or breastfeeding. (Lactating females must agree not to breast feed while taking lenalidomide)
* Patients seropositive for the human immunodeficiency virus (HIV).
* Prior organ transplant requiring immunosuppressive therapy.
* Patients who were previously exposed to higher doses of lenalidomide and who developed severe adverse events at higher doses that preclude incremental dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10-28 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hassoun, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Stamford Hospital, Stamford, Connecticut
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - North Shore LIJ, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 65 [47 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Population: A total of 10 patients were evaluable for the primary endpoint of response.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 10
participants
  Partial Response | 1
  Minor Response | 1
  Stable Disease | 7
  Progression of Disease | 1

2. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: All toxicities with a maximum grade and status of ≥ grade 2 will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: every 28 days before initiation of a new cycle through study completion until disease progression up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Blurred Vision (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT01463670/Prot_SAP_000.pdf